CLINICAL TRIAL: NCT04210297
Title: Development and Validation of an Noninvasive Model for Predicting High Risk Esophageal Varices in Cirrhosis
Status: Completed | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: Jinan Central Hospital (Other)
Responsible Party: Principal Investigator, Yanjing Gao, Clinical Professor, Qilu Hospital of Shandong University
Other Study IDs: LinMaxwell2018
Record Dates: First submitted 2019-12-15; First posted 2019-12-24 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Esophageal and Gastric Varices
Keywords: noninvasive; portal hypertension; radiomics
MeSH Terms: conditions — Esophageal and Gastric Varices; Hypertension, Portal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Training cohort: Training cohort consists of the cirrhotic patients who collected from January 2018 to December 2019 of Qilu Hospital retrospectively.
- Internal validation cohort: Internal validation cohort consists of the cirrhotic patients who enrolled from January 2020 of Qilu Hospital prospectively.
- External validation cohort: External validation cohort consists of the cirrhotic patients who enrolled from January 2020 in Jinan Central Hospital prospectively.

SUMMARY:
The aim of the study is to develop and validate a new noninvasive method based on routine examination during clinical practice for predicting high risk esophageal varices in cirrhosis.

DETAILED DESCRIPTION:
Portal hypertension is the main consequence of cirrhosis. Variceal bleeding is the principal and life-threatening complication of portal hypertension. Endoscopic screening is the golden standard to detect esophageal varices. However, endoscopy is limited by its invasiveness, cost and the discomfort it imposes on patients. With the goal of circumventing these disadvantages, we intend to develop an noninvasive method for predicting high risk esophageal varices.

ELIGIBILITY:
The inclusion criteria:

1. patients who were diagnosed with liver cirrhosis.
2. patients who underwent the abdominal contrast-enhanced CT examination.
3. patients who received endoscopic screening.
4. patients with written informed consent.

The exclusion criteria:

1. patients who previously underwent endoscopic therapy, transjugular intrahepatic portosystemic shunt (TIPS), splenectomy, partial splenic embolization (PSE), hepatectomy, balloon-occluded retrograde transvenous obliteration, or liver transplantation.
2. patients with liver cancer.
3. patients with severe ascites or hepatic encephalopathy.
4. lacks abdominal contrast-enhanced CT within 1 month of endoscopy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We queried the cirrhotic patients treated in Qilu Hospital Affiliated to Shandong University and Jinan Central Hospital Affiliated to Shandong University.
Sampling Method: Non-Probability Sample
Enrollment: 245 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Accuracy | through study completion, up to 2 years
  The golden standard is endoscopic examination.Compare the accuracy of the noninvasive model with the endoscopic examination.
sensitivity | through study completion, up to 2 years
  the sensitivity of predicting high risk esophageal varices of the noninvasive model.
specificity | through study completion, up to 2 years
  the specificity of predicting high risk esophageal varices of the noninvasive model.

CONTACTS AND LOCATIONS:
Overall Officials: Yanjing Gao, PhD.MD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Department of Gastroenterology,Qilu Hospital,Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin Y, Li L, Yu D, Liu Z, Zhang S, Wang Q, Li Y, Cheng B, Qiao J, Gao Y. A novel radiomics-platelet nomogram for the prediction of gastroesophageal varices needing treatment in cirrhotic patients. Hepatol Int. 2021 Aug;15(4):995-1005. doi: 10.1007/s12072-021-10208-4. Epub 2021 Jun 11. PMID 34115257